CLINICAL TRIAL: NCT04665440
Title: Variation of Salivary Oxytocin and Cortisol Levels in Premature Neonates and Their Mothers in Response to Multi-sensory Stimuli
Brief Title: Response of Preterm Infants to Multisensory Stimuli
Acronym: OXYVOICE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Prof. Olivier BAUD, MD-PhD, Professor, University Hospital, Geneva
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2020-00101
Record Dates: First submitted 2020-12-03; First posted 2020-12-11 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Mother-Infant Interaction
Keywords: neonates; oxytocin; late preterm; stress; family-centered intervention
MeSH Terms: interventions — Voice

STUDY DESIGN:
Intervention Model Description: prospective randomised crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Voice only then distraction (Other): First intervention: mother's voice without tactile stimuli Second intervention: mother's voice with tactile stimuli
  Interventions: Other: Voice alone; Other: Voice + tactile stimuli
- Distraction then voice only (Other): First intervention: mother's voice with tactile stimuli Second intervention: mother's voice without tactile stimuli
  Interventions: Other: Voice alone; Other: Voice + tactile stimuli

INTERVENTIONS:
Other: Voice alone — mother's voice without tactile stimuli
Other: Voice + tactile stimuli — mother's voice with tactile stimuli

SUMMARY:
The aim of this study is to measure the variation of oxytocin and cortisol levels in the saliva of premature neonates and their mother after sensorial stimuli.

DETAILED DESCRIPTION:
The aim of this study is to measure the variation of oxytocin and cortisol levels in the saliva of neonates with gestational age ranging from 32 to 34 completed weeks and in the saliva of their mothers. The measurements are taken before and after sensorial stimuli including mother voice exposure +/- tactile distraction for 10 minutes. The two interventions are performed between day 5 and day 12 after birth and 24 to 48 hours apart. Each child is randomised in a group depending on order of the two interventions.

Investigators hypothesize that an increase in the oxytocin/cortisol ratio will be occurred in neonates after hearing their mothers and that simultaneous tactile stimulation will mitigate that effect.

Concomitantly, the neonate's vital signs and his facial expressions are recorded during interventions. The mothers anxiety level is assessed PSS-NICU questionnaire given before the first and after the second intervention.

ELIGIBILITY:
Inclusion Criteria:

* Newborn gestational age 32 0/7 weeks to 34 6/7 weeks
* Born at university hospital Geneva
* French speaking parents
* Out of incubator
* Signed consent

Exclusion Criteria:

* Newborn with one of the above conditions:
* Congenital malformation
* intraventricular hemorrhage grade III or IV
* white matter abnormality
* anti-epileptic or sedative drugs
* altered consciousness level
* Infant requiring respiratory support
* psychiatric disorders in the mother or antenatal use of psychoactive drugs
* Bilateral absent otoacoustic emissions and/or auditory evoked potential
* Parents refusal to participate

Ages: 32 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Oxytocin/cortisol ratio | at baseline and 10 minutes after intervention
  Change in salivary oxytocin/cortisol ratio in response to the intervention

SECONDARY OUTCOMES:
Vital signs | at baseline, during and 10 minutes after intervention
  Change in heart rate and respiratory rate in response to the intervention
Facial expression analysis | at baseline, during and 10 minutes after intervention
  Response of neonate to intervention analysed by standardized neonatal facial coding system score, measured on video recording before, during and after the intervention
mother anxiety and mother infant bond | at baseline and 10 minutes after intervention
  Level of the mothers anxiety and her bond to the infant analyzed using NICU-PSS questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires Genève, Geneva, Switzerland

REFERENCES:
- [Background] Filippa M, Panza C, Ferrari F, Frassoldati R, Kuhn P, Balduzzi S, D'Amico R. Systematic review of maternal voice interventions demonstrates increased stability in preterm infants. Acta Paediatr. 2017 Aug;106(8):1220-1229. doi: 10.1111/apa.13832. Epub 2017 Apr 19. PMID 28378337
- [Background] Weber A, Harrison TM, Sinnott L, Shoben A, Steward D. Plasma and Urinary Oxytocin Trajectories in Extremely Premature Infants During NICU Hospitalization. Biol Res Nurs. 2017 Oct;19(5):549-558. doi: 10.1177/1099800417718266. Epub 2017 Jul 12. PMID 28699358
- [Background] Vittner D, McGrath J, Robinson J, Lawhon G, Cusson R, Eisenfeld L, Walsh S, Young E, Cong X. Increase in Oxytocin From Skin-to-Skin Contact Enhances Development of Parent-Infant Relationship. Biol Res Nurs. 2018 Jan;20(1):54-62. doi: 10.1177/1099800417735633. Epub 2017 Oct 11. PMID 29017336
- [Background] Zinni M, Colella M, Batista Novais AR, Baud O, Mairesse J. Modulating the Oxytocin System During the Perinatal Period: A New Strategy for Neuroprotection of the Immature Brain? Front Neurol. 2018 Apr 13;9:229. doi: 10.3389/fneur.2018.00229. eCollection 2018. PMID 29706926
- [Background] Lejeune F, Brand LA, Palama A, Parra J, Marcus L, Barisnikov K, Debillon T, Gentaz E, Berne-Audeoud F. Preterm infant showed better object handling skills in a neonatal intensive care unit during silence than with a recorded female voice. Acta Paediatr. 2019 Mar;108(3):460-467. doi: 10.1111/apa.14552. Epub 2018 Sep 21. PMID 30144160
- [Background] Kuhn P, Sizun J, Casper C; GREEN study group from the French Neonatal Society. Recommendations on the environment for hospitalised newborn infants from the French neonatal society: rationale, methods and first recommendation on neonatal intensive care unit design. Acta Paediatr. 2018 Nov;107(11):1860-1866. doi: 10.1111/apa.14501. Epub 2018 Aug 13. PMID 30025190